CLINICAL TRIAL: NCT00936273
Title: Screening for Sleep Apnea Using Home Recording of the Double Loop Gain as a Measure of Periodic Breathing
Brief Title: Sleep Apnea and Periodic Breathing
Acronym: DLI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Dr. J.G. van den Aardweg, MD, Medical Center Alkmaar
Other Study IDs: Double loop gain MCA 2009
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Sleep Apnea Syndrome
Keywords: Sleep apnea syndrome; SAS; double loop gain; DLI; double loop index; periodic breathing; polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected sleep apnea syndrome: Outpatients with suspected sleep apnea syndrome, age > 18 year

SUMMARY:
The purpose of this study is to determine the double loop index (DLI) threshold with optimal sensitivity and specificity. The investigators hypothesize that the DLI gives a better reflection of the pathophysiology of the disease than the apnea-hypopnea-index (AHI).

DETAILED DESCRIPTION:
Sleep apnea syndrome (SAS) is characterized by repetitive events of apnea and hypopnea. These events are often part of a periodic breathing pattern, in which relative hyperventilation is followed by apnea or hypopnea.

Recently the investigators described the 'double-loop gain' of the respiratory control system as a measure of periodic breathing. This is a frequency-dependent variable which describes 1) the tendency of the respiratory system to oscillate at a given frequency and 2) the degree to which the relation between oscillations in ventilation and oscillations in arterial blood gas values is linear. The underlying hypothesis is that periodic breathing results from negative feedback regulation of arterial O2 and CO2 pressure through the chemoreflexes. The double-loop gain describes the gain in the negative feedback loop under the assumption that accidental changes occur in both ventilation and arterial blood gas pressures. A simple version of the double-loop gain is derived from nasal pressure changes and arterial O2 saturation. From all-night recordings, the 'double-loop index' (DLI) can be derived, which is determined by the time during which the double-loop gain exceeds a given threshold.

Currently, the presence of sleep-apnea is determined by the apnea-hypopnea index (AHI), using in-hospital sleep recording. With a growing number of referrals, waiting lists for sleep registration are emerging. Screening for SAS using home-measurement of nasal pressure and SaO2 seems to be a good alternative. The investigators hypothesize that the DLI derived from these signals gives a better reflection of the pathophysiology of the disease than the AHI. As a result, the investigators expect that the DLI improves the distinction between healthy and diseased subjects in comparison to the simple counting of apneas and hypopneas. This is reflected in a higher area under the ROC curve, which describes the sensitivity and specificity of the test.

ELIGIBILITY:
Inclusion Criteria:

* Suspected sleep apnea syndrome
* > 18 yr
* Outpatient
* Able and willing to use the necessary equipment for registration of nasal pressure and O2 saturation at home

Exclusion Criteria:

* hospitalized patients
* < 18 yr
* Not able to use the necessary equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients suspected for sleep apnea syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
To determine DLI threshold with optimal sensitivity and specificity. The DLI threshold is the DLI value above which the test is considered positive. The optimal DLI threshold will be taken as the value that gives the highest area under the ROC curve. | 1 year

SECONDARY OUTCOMES:
To test the hypothesis that the sensitivity and specificity of the screening are higher when the DLI is used instead of the AHI | 1 year
To assess the repeatability of the DLI using home and in-hospital recordings of nasal pressure and saturation (SaO2). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J.G. van den Aardweg, dr, Study Director — Medical Center Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, Wilhelminalaan 12, Netherlands